CLINICAL TRIAL: NCT06297928
Title: Metabolomics and Bariatric Surgery in Patients With Metabolically Unhealthy Obesity: Advancing Precision Medicine for the Treatment of Obesity
Brief Title: Metabolomics and Bariatric Surgery in Patients With Metabolically Unhealthy Obesity
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/11238/I
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid; Obesity, Metabolically Benign
Keywords: bariatric surgery; Metabolically Unhealthy Obesity; metabolomics; Clinical obesity; subclinical obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity, Metabolically Benign

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: baratric surgery — Participants in this study will undergo bariatric surgery, either gastric bypass or sleeve gastrectomy, based on clinical criteria and consensus from a multidisciplinary team.

SUMMARY:
The goal of this observational study is to investigate metabolic changes in individuals undergoing bariatric surgery, specifically focusing on those with obesity and varying metabolic health statuses. The main questions it aims to answer are:

* Can metabolic markers predict the transition from metabolically unhealthy obesity to metabolically healthy obesity after bariatric surgery?
* How do metabolic profiles change in individuals with metabolically healthy obesity after bariatric surgery?
* What are the metabolic differences between individuals with metabolically healthy and unhealthy obesity before and after bariatric surgery?

Participants will undergo routine evaluations and blood tests before and after bariatric surgery. These tests will include assessments of metabolic health markers and sampling of blood plasma for metabolomic analysis. The study will study changes in metabolic profiles between individuals who transition to metabolically healthy obesity and those who remain metabolically unhealthy after surgery.

In January 2025, a new definition of clinical obesity was proposed by the Lancet Commission, focusing on organ/system dysfunction induced by excess adiposity. In response, this study has expanded its objectives to assess the prevalence, predictors, and metabolomic correlates of clinical obesity and its remission after bariatric surgery.

DETAILED DESCRIPTION:
This is a prospective observational study conducted at the bariatric surgery unit. Patients undergo routine assessments and preoperative evaluations by a multidisciplinary team including surgeons, endocrinologists, nutritionists, psychologists, psychiatrists, and anesthesiologists. Clinical evaluations include physical examinations and laboratory tests to detect cardiometabolic comorbidities before surgery. The two bariatric surgery techniques performed in this center are gastric bypass and vertical gastrectomy. The choice of technique is based on clinical criteria and consensus of the multidisciplinary team. After surgery, patients are evaluated at 3, 6, and 12 months through anthropometry, blood pressure measurements, smoking habits assessment, and routine blood analysis. Patients are invited to participate in the OBEMAR registry during the preoperative period. With informed consent, patients authorize the collection of serum and plasma samples at each visit for scientific purposes. Participation in the study does not entail additional visits or procedures beyond standard clinical practice and participation in the OBEMAR registry.

Metabolically Health Status Criteria:

Health status will be defined according to the criteria used by Wildman et al. in the NHANES 1999-2004 study, excluding C-reactive protein measurement. Patients will be classified as metabolically healthy obese (OMS) if they have only one or none of the cardiometabolic factors. Patients with two or more risk factors will be categorized as metabolically unhealthy obese (OME). This classification will be performed before and one year after surgery.

Metabolomics The study will analyze various metabolites related to amino acid metabolism, energy metabolism, and lipid profile. These metabolites will provide insights into metabolic changes before and after bariatric surgery. Specifically, the study will focus on branched-chain amino acids (BCAA), aromatic amino acids (AAA), energy metabolites, and lipid species.

Sample size and origin To ensure statistical power, a sample size calculation was performed based on the anticipated distribution of patients transitioning to metabolically healthy obesity (OMS) or maintaining metabolically unhealthy obesity (OME) status after surgery. It is estimated that 84.4% of patients will transition to OMS, while the remaining 15.6% will remain OME after surgery. Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-tailed test, a minimum of 19 subjects in the OME group and 102 in the OMS group are required to detect a difference of 25% or more in the selected metabolites. Assuming a common standard deviation of 35% for these metabolites, a total of 145 patients need to be included to ensure that 121 meet OME criteria before surgery.

Patients for this study will be sourced from the OBEMAR registry, which comprises individuals who have undergone bariatric surgery at the Hospital del Mar. A portion of the patients included in this registry already have sufficient clinical information to classify them as OMS or OME, and their biological samples are stored in a biobank. As of February 2023, complete clinical data and pre- and post-operative samples are available for 70 patients. With approximately 100 surgeries performed annually in our unit, it is anticipated that the desired sample size will be attained by July 2025.

In January 2025, an international expert commission published a new definition of clinical obesity in The Lancet Diabetes & Endocrinology, shifting the paradigm from traditional risk-based classifications (such as the metabolically healthy/unhealthy obesity concept) to a functional definition based on organ and system-level dysfunctions attributable to excess adiposity. This new definition aims to set a precedent in public health policies, pharmacological treatment indications, and the clinical organization of obesity care. However, it has sparked considerable debate among experts and scientific societies regarding its impact, applicability, and clinical validity.

Given this context, it is essential to generate new knowledge around this concept. Although this study was initially designed to explore a specific metabolic phenotype (metabolically healthy obesity), it now represents a unique opportunity to evaluate the prevalence, predictors, and mechanisms associated with clinical obesity and its remission after bariatric surgery. This adaptation aligns with the research priorities outlined by the expert commission, which emphasize the need to:

Identify biomarkers and/or anthropometric criteria to improve the diagnosis and prognostic stratification of clinical obesity.

Evaluate the efficacy of current anti-obesity interventions in terms of remission or improvement of clinical obesity-not just weight loss or reduced risk of comorbidities.

Understand the degree of weight loss necessary to induce meaningful clinical improvement.

Advance the prevention and treatment of clinical and pre-clinical obesity using a precision medicine approach.

Incorporating these goals, this study will provide valuable insights into how bariatric surgery and metabolomic profiles relate to the new framework of clinical obesity, potentially influencing future therapeutic strategies and clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing bariatric surgery at the Hospital del Mar in Barcelona. Criteria for bariatric surgery are:

* Ages between 18 and 60 years.
* Body Mass Index (BMI) equal to or greater than 40, or equal to or greater than 35 kg/m2 with at least one obesity-related comorbidity (type 2 diabetes mellitus, hypertension, dyslipidemia, obstructive sleep apnea syndrome).
* Previous failure with conventional treatment involving diet and exercise.

Exclusion Criteria:

* History of previous bariatric surgery.
* Presence of severe psychiatric disorders, severe eating disorders, alcohol or drug abuse.
* Contraindications for major abdominal surgery, active gastric ulcer, severe liver disease.

Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The study population will consist of patients who have undergone bariatric surgery at the Hospital del Mar in Barcelona and meet the aforementioned inclusion criteria. These patients will be consecutively selected and must agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Identification of Metabolic Signatures Using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) Analysis Predicting Transition from Metabolically Unhealthy Obesity (MUO) to Metabolically Healthy Obesity (MHO) Status | The transition from MUO to MHO status will be assessed at one year after bariatric surgery.
  The primary objective of this study is to identify metabolic signatures present in patients with metabolically unhealthy obesity (MUO) before bariatric surgery, which can predict the transition to metabolically healthy obesity (MHO) status one year after the intervention.
  For patients meeting the criteria for MUO before surgery, a comparison will be made between those who remain MUO at 12 months post-intervention and those who transition to MHO. The baseline metabolomic profile, measured using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS), will be compared between these groups

SECONDARY OUTCOMES:
Comparison of Metabolomic Changes Using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) between Patients with Persistent Metabolically Unhealthy Obesity (MUO) and Those Transitioning to Metabolically Healthy Obesity (MHO) Status | Metabolomic changes will be assessed at 3 and 12 months after bariatric surgery
  The secondary objective of this study is to compare the changes in metabolomic profiles between patients with persistent metabolically unhealthy obesity (MUO) and those who transition to metabolically healthy obesity (MHO) status one year after bariatric surgery. We aim to elucidate the metabolic pathways associated with successful metabolic health improvement following surgery.
Comparison of Baseline Metabolomic Profile and Its Evolution Using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) after Surgery between Patients with Metabolically Healthy Obesity (MHO) and Metabolically Unhealthy Obesity (MUO) | Baseline metabolomic profiling will be conducted before surgery. The evolution of metabolomic profiles will be assessed at 3 and 12 months post-surgery.
  This study aims to compare the baseline metabolomic profiles and their evolution after surgery between patients with metabolically healthy obesity (MHO) and metabolically unhealthy obesity (MUO) using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) analysis. We will compare the metabolic signatures of patients classified as MHO and MUO before bariatric surgery. Specifically, we will compare the baseline metabolomic profiles and the changes in the metabolome at 3 and 12 months post-surgery. This analysis will provide insights into the metabolic mechanisms underlying metabolic health improvement after bariatric surgery.
Prevalence of Clinical Obesity at Baseline and Rate of Transition to Subclinical Obesity One Year After Bariatric Surgery | Assessed at baseline and at 12 months after bariatric surgery.
  This objective seeks to quantify the prevalence of clinical obesity in patients undergoing bariatric surgery according to the criteria established by the 2025 Lancet Commission. It will also assess the rate of transition from clinical to subclinical obesity status at 12 months postoperatively.
Identification of Metabolic Signatures Using LC-MS/MS Predicting Transition from Clinical Obesity to Subclinical Obesity Status | Metabolomic changes will be assessed at 3 and 12 months after bariatric surgery.
  This secondary objective aims to identify metabolomic signatures present in patients with clinical obesity (as defined by the 2025 Lancet Commission) before bariatric surgery, which can predict the transition to subclinical obesity status one year after the intervention. Among patients classified as having clinical obesity preoperatively, comparisons will be made between those who remain in clinical obesity status and those who transition to subclinical obesity at 12 months. Baseline metabolomic profiles will be measured using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) and compared between these groups.
Comparison of Metabolomic Changes Using Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) Between Patients With Persistent Clinical Obesity and Those Transitioning to Subclinical Obesity | Baseline, 3 months, and 12 months after bariatric surgery.
  This objective aims to compare the metabolomic changes over time in patients classified as having clinical obesity before bariatric surgery, based on the 2025 Lancet Commission definition. Patients who maintain clinical obesity at 12 months postoperatively will be compared with those who transition to subclinical obesity. Longitudinal changes in metabolomic profiles, measured by LC-MS/MS at baseline, 3 months, and 12 months, will be analyzed to identify metabolic pathways associated with organ/system recovery and clinical improvement after bariatric surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goday A, Benaiges D, Parri A, Ramon JM, Flores-Le Roux JA, Pedro Botet J; Obemar Group. Can bariatric surgery improve cardiovascular risk factors in the metabolically healthy but morbidly obese patient? Surg Obes Relat Dis. 2014 Sep-Oct;10(5):871-6. doi: 10.1016/j.soard.2014.04.022. Epub 2014 May 2. PMID 25282193
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Dang JT, Mocanu V, Park H, Laffin M, Tran C, Hotte N, Karmali S, Birch DW, Madsen K. Ileal microbial shifts after Roux-en-Y gastric bypass orchestrate changes in glucose metabolism through modulation of bile acids and L-cell adaptation. Sci Rep. 2021 Dec 10;11(1):23813. doi: 10.1038/s41598-021-03396-4. PMID 34893681
- [Background] de Hollanda A, Ruiz T, Jimenez A, Flores L, Lacy A, Vidal J. Patterns of Weight Loss Response Following Gastric Bypass and Sleeve Gastrectomy. Obes Surg. 2015 Jul;25(7):1177-83. doi: 10.1007/s11695-014-1512-7. PMID 25421881
- [Background] Rawlins ML, Teel D 2nd, Hedgcorth K, Maguire JP. Revision of Roux-en-Y gastric bypass to distal bypass for failed weight loss. Surg Obes Relat Dis. 2011 Jan-Feb;7(1):45-9. doi: 10.1016/j.soard.2010.08.013. Epub 2010 Sep 15. PMID 21111688
- [Background] Fultang J, Chinaka U, Rankin J, Bakhshi A, Ali A. Preoperative Bariatric Surgery Predictors of Type 2 Diabetes Remission. J Obes Metab Syndr. 2021 Jun 30;30(2):104-114. doi: 10.7570/jomes20084. PMID 33436532
- [Background] Kim EY. Definition, Mechanisms and Predictors of Weight Loss Failure After Bariatric Surgery. J Metab Bariatr Surg. 2022 Dec;11(2):39-48. doi: 10.17476/jmbs.2022.11.2.39. Epub 2023 Feb 3. PMID 36926678
- [Background] Sun YV, Hu YJ. Integrative Analysis of Multi-omics Data for Discovery and Functional Studies of Complex Human Diseases. Adv Genet. 2016;93:147-90. doi: 10.1016/bs.adgen.2015.11.004. Epub 2016 Jan 25. PMID 26915271
- [Background] Olivier M, Asmis R, Hawkins GA, Howard TD, Cox LA. The Need for Multi-Omics Biomarker Signatures in Precision Medicine. Int J Mol Sci. 2019 Sep 26;20(19):4781. doi: 10.3390/ijms20194781. PMID 31561483
- [Background] Vaz M, Pereira SS, Monteiro MP. Metabolomic signatures after bariatric surgery - a systematic review. Rev Endocr Metab Disord. 2022 Jun;23(3):503-519. doi: 10.1007/s11154-021-09695-5. Epub 2021 Dec 2. PMID 34855133
- [Background] Arora T, Velagapudi V, Pournaras DJ, Welbourn R, le Roux CW, Oresic M, Backhed F. Roux-en-Y Gastric Bypass Surgery Induces Early Plasma Metabolomic and Lipidomic Alterations in Humans Associated with Diabetes Remission. PLoS One. 2015 May 6;10(5):e0126401. doi: 10.1371/journal.pone.0126401. eCollection 2015. PMID 25946120
- [Background] Kwon Y, Jang M, Lee Y, Ha J, Park S. Metabolomic Analysis of the Improvements in Insulin Secretion and Resistance After Sleeve Gastrectomy: Implications of the Novel Biomarkers. Obes Surg. 2021 Jan;31(1):43-52. doi: 10.1007/s11695-020-04925-2. Epub 2020 Aug 19. PMID 32815103
- [Background] Stefan N, Haring HU, Hu FB, Schulze MB. Metabolically healthy obesity: epidemiology, mechanisms, and clinical implications. Lancet Diabetes Endocrinol. 2013 Oct;1(2):152-62. doi: 10.1016/S2213-8587(13)70062-7. Epub 2013 Aug 30. PMID 24622321
- [Background] Caleyachetty R, Thomas GN, Toulis KA, Mohammed N, Gokhale KM, Balachandran K, Nirantharakumar K. Metabolically Healthy Obese and Incident Cardiovascular Disease Events Among 3.5 Million Men and Women. J Am Coll Cardiol. 2017 Sep 19;70(12):1429-1437. doi: 10.1016/j.jacc.2017.07.763. PMID 28911506
- [Background] Soriguer F, Gutierrez-Repiso C, Rubio-Martin E, Garcia-Fuentes E, Almaraz MC, Colomo N, Esteva de Antonio I, de Adana MS, Chaves FJ, Morcillo S, Valdes S, Rojo-Martinez G. Metabolically healthy but obese, a matter of time? Findings from the prospective Pizarra study. J Clin Endocrinol Metab. 2013 Jun;98(6):2318-25. doi: 10.1210/jc.2012-4253. Epub 2013 Apr 4. PMID 23559087
- [Background] Bluher M. Are there still healthy obese patients? Curr Opin Endocrinol Diabetes Obes. 2012 Oct;19(5):341-6. doi: 10.1097/MED.0b013e328357f0a3. PMID 22895358
- [Background] Goday A, Julia H, de Vargas-Machuca A, Pedro-Botet J, Benavente S, Ramon JM, Pera M, Casajoana A, Villatoro M, Fontane L, Bisbe M, Climent E, Castaner O, Flores Le Roux JA, Benaiges D. Bariatric surgery improves metabolic and nonalcoholic fatty liver disease markers in metabolically healthy patients with morbid obesity at 5 years. Surg Obes Relat Dis. 2021 Dec;17(12):2047-2053. doi: 10.1016/j.soard.2021.07.021. Epub 2021 Aug 12. PMID 34509375